CLINICAL TRIAL: NCT03065725
Title: Is Late FDG-PET/CT Imaging Better Than Early FDG-PET/CT Imaging to Distinguish Between Malign and Inflammatory Changes in Lymph Nodes in Patients With Muscle Invasive Bladder Cancer Scheduled for Radical Cystectomy?
Brief Title: Early Versus Late FDG-PET/CT in Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Jørgen Bjerggaard Jensen (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: PETCT2
Record Dates: First submitted 2017-02-10; First posted 2017-02-28 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: late FDG — In addition to regular FDG-PET/CT 60 minutes post injection, an extra scan 180 minutes post injection is made.

SUMMARY:
The aim of this study is to examine if late FDG-PET/CT images after intravenous FDG injection has a higher sensitivity and specificity in detecting local lymph node metastases in patients with muscle invasive BC than FDG-PET/CT images 60 minutes after FDG injection. The latter procedure has been used routinely until now.

DETAILED DESCRIPTION:
Background: Approximately 900 patients are diagnosed with invasive bladder cancer (BC) in Denmark each year. Approximately 50% are diagnosed with non-muscle invasive BC (T1) and approximately 50% are diagnosed with a muscle invasive BC (T2-4). Male-female ratio is 75% - 25% and the median age among all diagnosed patients at time of diagnose is 73 years (range 32 - 98) (national data from September 1st 2014 to august 31st 2015).1 One third of all diagnosed patients will be treated with surgical removal of the urinary bladder, radical cystectomy (RC). Additional 14% will receive curative intended radiotherapy. At the Department of Urology, Aarhus University Hospital, approximately 120 patients will be treated with RC due to BC every year.

2-[18F]-Fluoro-2-deoxy-D-glucose (FDG) - positron emission tomography (PET) /computed tomography (CT) is standard for primary staging at Aarhus University Hospital, Denmark, when evaluating patients with muscle invasive BC before radical curative intended treatment.

Evaluation of disease stage is done by investigation for lymph node metastasis and non-local metastases separately.

FDG is a radioactively marked glucose analogue used as a tracer for cells with high glucose uptake. The uptake of glucose in most malignant cells are much greater than the glucose uptake in normal cells. Because of this, FDG can be used as a tracer in the diagnosis of cancers and hereby also BC. However, FDG is not a cancer specific tracer. Cells of the immune system like neutrophil leucocytes, macrophages and lymphocytes also have high glucose uptake and thus, high FDG uptake. Being a glucose analogue, the uptake of FDG in the cells is similar to the uptake of glucose by, the transport protein GLUT-1. Inside the cells FDG is phosphorylated into FDG-6-phosphate by the enzyme hexokinase. FDG-6-phosphate is not metabolized further and is trapped inside the cells. Malignant cells have a tendency to up-regulate both GLUT-1 and hexokinase which results in increase FDG uptake in cancer cells. Hereby optimizing imagine of primary tumour and possible metastasis but also possible inflammatory changes.

After intravenous injection of FDG, the distribution of FDG in the body can be visualized by performing a PET-scan. FDG-PET has a high sensitivity in detecting even small malignant changes but is not very specific to show the anatomical localization of these changes. Thus, the FDG-PET is combined with a CT-scan, which has a high sensitivity in anatomical localization. Hybrid PET/CT scanners are now widely used for imaging.

International studies have shown that FDG-PET/CT is superior to CT and magnetic resonance (MR) alone in detecting lymph node metastasis in patients with BC.2,3

Aim: The aim of this study is to examine if late FDG-PET/CT images after intravenous FDG injection has a higher sensitivity and specificity in detecting local lymph node metastases in patients with muscle invasive BC than FDG-PET/CT images 60 minutes after FDG injection. The latter procedure has been routinely until now.

Hypothesis: FDG-PET/CT after 180 minutes post injection (PI) will have a higher specificity than FDG-PET/CT after 60 minutes PI regarding differentiation between local lymph node metastasis and benign inflammatory changes in local lymph nodes when evaluating patients with muscle invasive BC before radical treatment.

Method: 200 consecutive patients diagnosed with muscle invasive BC and candidate for radical cystectomy will be examined with an FDG-PET/CT scan as primary staging for evaluation of local lymph node metastasis and distant metastasis. In our standard procedure, the patient is given intravenous FDG and will rest for 30 minutes and after 60 minutes a PET/CT-scan will be performed. The PET/CT scan will be performed over the course of 25-40 minutes. In this study, the included patients will have an additional PET/CT (low dose)-scan of the pelvic area performed 180 minutes PI.

The FDG-PET/CT scans will be evaluated by a experienced specialist in nuclear medicine together with a experienced specialist in radiology. SUVmax values of regional lymph nodes on early and late images will be compared with histology of removed lymph nodes.

Lymph node dissection during cystectomy will be performed according to an extended template with the aortic bifurcation as the proximal limit. Lymph nodes or lymph node packages that are FDG-positive on the preoperative PET/CT will be send marked separately for pathological evaluation if possible. All dissected lymph nodes will undergo pathological evaluation.

Histological evaluation will be performed by a specialist from the Institute of Pathology on histological tissue either from a needle biopsy or from dissected lymph nodes at the time of cystectomy.

The study will take place between the 1th of January 2017 and until a total of 100 patients are included, which is expected to be by the end of 2018.

Ethical aspects:

Patients included in this study will only receive small additional radiation dose (1-1 1/2 mSv) due to the extra low dose CT of the pelvic area. The patients will not receive further radiation dose from FDG. The patients will have a longer stay at The Department of Nuclear & PET Center due to the extra PET/CT scan 2 hours after the first PET/CT scan. Duration of the extra scan of the pelvic area is 6-8 min. The radiation dose from the standard FDG PET/CT in bladder cancer is 18-28 mSv.

The regional ethics committee of Central Denmark Region was notified of the study. They considered this to be quality assurance and hence had no objections to the performance of the study.

After one year inclusion preliminary results will be evaluated. It is expected that 50 patients will be included by this time.

Perspectives: As of today it is common practice that all patients who are found possibly suitable for cystectomy due to BC will get an FDG-PET/CT performed prior to treatment to evaluate their disease stage. The sensitivity for FDG-PET/CT in detecting malignant local lymph nodes is high. The specificity, however, is invert proportional depending on SUVmax cut-off. If a method of improving the specificity could be found this would mean a significant difference for some of the patients who may get a better treatment due to their BC with lower mortality over time.

If the study finds that PET scan 180 minutes after FDG injection has a higher specificity in detecting malign local lymph nodes in patients with BC than PET scan after 60 minutes, we will change our procedure according to this. As a consequence, it will be better to evaluate the BC patients prior to potential curative treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with BC who are candidates for cystectomy and undergo cystectomy with lymph node dissection or have a needle biopsy of at least one FDG-PET/CT local lymph node suspected for malignancy following the FDG-PET/CT due to their BC.

Exclusion criteria:

* Patients who have received chemotherapy, including neoadjuvant chemotherapy, in the timespan between the FDG-PET/CT and the needle biopsy or the lymph node dissection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bladder cancer scheduled for cystectomy
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Patient with preoperatively detection of metastasis in lymph nodes | baseline
  Number of patients with metastasis proven in lymph nodes by preoperative PET/CT

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hospital of West Jutland, Holstebro, Danmark
  - Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No